CLINICAL TRIAL: NCT00577109
Title: An Open Label Study to Assess the Effect of FOLFIRI Plus Avastin and Cetuximab on Progression-free Survival in Patients With Previously Untreated Metastatic Colorectal Cancer.
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Chemotherapy in Patients With Previously Untreated Metastatic Colorectal Cancer.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled before patient enrollment
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20452
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Leucovorin; Cetuximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Irinotecan; Drug: Leucovorin; Drug: 5 FU; Drug: Cetuximab

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5mg/kg iv on day 1 of each 2 week cycle
Drug: Irinotecan — 180mg/m2 iv on day 1 of each 2 week cycle
Drug: Leucovorin — 200mg/m2 iv on day 1 of each 2 week cycle
Drug: 5 FU — 400mg/m2 iv on day 1 of each 2 week cycle
Drug: Cetuximab — Loading dose of 400mg/m2 iv followed by 250mg/m2 iv on day 3 of each 2 week cycle

SUMMARY:
This single arm study will assess the efficacy and safety of a combination of modified FOLFIRI (irinotecan, 5-FU and leucovirin), Avastin and cetuximab in patients with previously untreated metastatic colorectal cancer. Patients will receive modified FOLFIRI (irinotecan 180mg/m2 iv, leucovirin 200mg/m2 iv, and 5-FU 400mg/m2 iv) on day 1 of each 2 week cycle, in combination with Avastin (5mg/kg iv on day 1 of each cycle) and cetuximab (loading dose of 400mg/m2 followed by 250mg/m2 on day 3 of each cycle). The anticipated time on study treatment is until disease progression or unacceptable toxicity, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* colorectal cancer;
* advanced or recurrent disease;
* >=1 measurable lesion;
* >=6 months since prior adjuvant therapy, and >=4 weeks since prior radiotherapy.

Exclusion Criteria:

* previous treatment for colorectal cancer;
* significant history of cardiac disease in past 6 months;
* other invasive malignancy within past 5 years, except for nonmelanoma skin cancer, and successfully treated cervical or prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12 (Estimated); Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 months

SECONDARY OUTCOMES:
Objective response rate, rate of resection of hepatic metastases, overall survival. | Event driven
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Brazil (3):
  - Salvador
  - São Paulo
  - Sorocaba